CLINICAL TRIAL: NCT02227186
Title: Study of Effectiveness of a School-located Influenza Vaccination Program in Raising Influenza Vaccination Rates
Brief Title: Efficacy Study of School-located Influenza Vaccination Clinics to Increase Influenza Vaccination Rates in Monroe County, New York
Acronym: SKIPP RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Peter G Szilagyi, MD MPH, Professor and Vice-Chair for Clinical Research, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 5R18HS021163 (AHRQ); 5R18HS021163 (AHRQ)
Record Dates: First submitted 2014-08-25; First posted 2014-08-28 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Childhood Influenza Vaccination; School-located Influenza Vaccination
Keywords: Influenza vaccination rates

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control arm (No Intervention): No school-located influenza vaccination clinic
- School-located influenza vaccination clinics (Experimental): School-located influenza vaccination clinics
  Interventions: Other: School-located Influenza Vaccination Clinic

INTERVENTIONS:
Other: School-located Influenza Vaccination Clinic — Children in the intervention arm are enrolled in schools in Monroe County, NY that are offering school-located influenza vaccination clinics during school hours
  Arms: School-located influenza vaccination clinics

SUMMARY:
Children in schools in which influenza vaccination clinics are held during school hours will have higher rates of influenza vaccination than children in control schools (no school-located clinics offered)

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in participating, randomized school

Exclusion Criteria:

* None

Ages: 4 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20461 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2015-07-31 (Actual); Study Completion 2015-07-31 (Actual)

PRIMARY OUTCOMES:
Influenza vaccination status | Within one year
  Vaccination status for the 2014/2015 influenza season will be assessed. The vaccination date will be recorded, as well as the provider name, to determine whether vaccine was received at the school-located influenza clinic

CONTACTS AND LOCATIONS:
Overall Officials: Peter Szilagyi, MPH, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester School of Medicine and Dentistry, Rochester, New York, United States

REFERENCES:
- [Derived] Yoo BK, Schaffer SJ, Humiston SG, Rand CM, Goldstein NPN, Albertin CS, Concannon C, Szilagyi PG. Cost effectiveness of school-located influenza vaccination programs for elementary and secondary school children. BMC Health Serv Res. 2019 Jun 24;19(1):407. doi: 10.1186/s12913-019-4228-5. PMID 31234842
- [Derived] Schaffer SJ, Rand CM, Humiston SG, Concannon C, Hightower AD, Albertin C, Szilagyi PG. Practical considerations in developing a successful school-located influenza vaccination (SLIV) program. Vaccine. 2019 Apr 10;37(16):2171-2173. doi: 10.1016/j.vaccine.2019.01.088. Epub 2019 Mar 13. No abstract available. PMID 30878250
- [Derived] Szilagyi PG, Schaffer S, Rand CM, Goldstein NPN, Younge M, Mendoza M, Albertin CS, Concannon C, Graupman E, Hightower AD, Yoo BK, Humiston SG. Text Message Reminders for Child Influenza Vaccination in the Setting of School-Located Influenza Vaccination: A Randomized Clinical Trial. Clin Pediatr (Phila). 2019 Apr;58(4):428-436. doi: 10.1177/0009922818821878. Epub 2019 Jan 2. PMID 30600690
- [Derived] Szilagyi PG, Schaffer S, Rand CM, Goldstein NPN, Vincelli P, Hightower AD, Younge M, Eagan A, Blumkin A, Albertin CS, DiBitetto K, Yoo BK, Humiston SG. School-located Influenza Vaccinations for Adolescents: A Randomized Controlled Trial. J Adolesc Health. 2018 Feb;62(2):157-163. doi: 10.1016/j.jadohealth.2017.09.021. Epub 2017 Dec 13. PMID 29248390
- [Derived] Szilagyi PG, Schaffer S, Rand CM, Vincelli P, Eagan A, Goldstein NP, Hightower AD, Younge M, Blumkin A, Albertin CS, Yoo BK, Humiston SG. School-Located Influenza Vaccinations: A Randomized Trial. Pediatrics. 2016 Nov;138(5):e20161746. doi: 10.1542/peds.2016-1746. PMID 27940785